CLINICAL TRIAL: NCT01371851
Title: Clinical Efficacy of Doxazosin for Psychostimulant Dependence
Brief Title: Doxazosin for Psychostimulant Dependence
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2-P50-DA018197-DoxMeth; 2P50DA018197 (NIH)
Record Dates: First submitted 2011-06-09; First posted 2011-06-13 (Estimated); Results first posted 2015-07-27 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Methamphetamine or Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Doxazosin (Experimental): Doxazosin extended release will be administered initially at 4 mg/day. On day 8 the dose is increased to 8 mg/day and the participant is maintained on the study until the end of the trial.
  Interventions: Drug: Doxazosin extended release
- Placebo (Placebo Comparator): Participants will be maintained on placebo (cellulose) throughout the trial.
  Interventions: Drug: Doxazosin extended release

INTERVENTIONS:
Drug: Doxazosin extended release — initially maintained on doxazosin extended release 4 mg once a day for 7 days, then the dose is increased to 8 mg once per day for the duration of the trial.

SUMMARY:
Psychostimulant dependence is a major public health problem and no medications have been shown to be very effective in treating this disorder. Thus, the investigators wish to study whether a blood pressure drug thought to reduce drug craving through its interaction at particular adrenergic receptors - doxazosin - can dredge cocaine use relative to placebo in psychostimulant dependent participants enrolled in an 8-week, randomized, double blind, placebo-controlled outpatient clinical trial. Our hypothesis is that doxazosin will reduce cocaine use relative to placebo in psychostimulant dependent participants.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years old
* Methamphetamine OR cocaine dependence, as assessed by the substance abuse section of the Structured Clinical Interview for DSM-IV.
* At least weekly self-reported methamphetamine OR cocaine use during a preceding three month period
* Urine toxicology screen positive for methamphetamine or methamphetamine metabolite OR cocaine or cocaine metabolite
* Women of childbearing age must have a negative pregnancy test, agree to adequate contraception to prevent pregnancy during the study, agree to monthly pregnancy testing and not be nursing

Exclusion Criteria:

* Suicide attempts within the past 12 months or suicidal ideations or psychotic symptoms in the past 6 months as determined by a study physician.
* Current opioid, alcohol or sedative physical dependence or dependence on both cocaine and methamphetamine
* Major cardiovascular disorder that contraindicates study participation (e.g., history of myocardial infarction, stroke, congestive heart failure, cardiac arrhythmia, significant hypertension [i.e., >170 SBP or >110 DBP] or an unstable medical condition (e.g., untreated bacterial infection) as determined by the study physician.
* Any history or evidence suggestive of seizure disorder or brain injury
* Subjects needing or planning cataract surgery.
* History of schizophrenia, major depression, or bipolar type I disorder
* Organic brain disease or dementia assessed by physician
* Use of medications that would be expected to have major interaction with doxazosin (e.g. atanazavir, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, or voriconazole or any other potent 3A4 inhibitor.,)
* Any previous medically adverse reaction to methamphetamine or cocaine, including loss of consciousness, chest pain, or epileptic seizure
* Medical contraindication to receiving doxazosin (e.g. liver problems or allergies to other to other quinazolines such as prazosin or terazosin)
* Severe gastrointestinal disorder as determined by physician
* Liver function tests (i.e., liver enzymes) greater than three times normal levels
* Systolic blood pressure > 170 mmHg or < 90 mmHg, diastolic blood pressure > 110 mmHg or < 60 mmHg, or heart rate of > 110 beats/min or < 55 beats/min.
* Supine blood pressure of 100/65 mm Hg or lower, a seated blood pressure of 90/60 mm Hg or lower, or an orthostatic change of >20mm Hg systolic or 10 mm Hg diastolic on standing.
* Have evidence of untreated or unstable medical illness including: neuroendocrine, autoimmune, renal, hepatic, or active infectious disease
* Have symptomatic HIV or are taking antiretroviral medication
* Have asthma or currently use theophylline or other sympathomimetics
* Participants with estimated glomerular filtration rate < 30 ml/min.
* Pregnant or nursing female

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2011-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UAMS Psychiatric Research Institute, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Doxazosin | Placebo
Started | 11 (Eligible participants who showed up on day 1 of week 1 and received at least one dose of study med.) | 11 (Eligible participants who showed up on day 1 of week 1 and received at least one dose of study med.)
Completed | 3 | 2
Not Completed | 8 | 9
Not completed — Lost to Follow-up | 5 | 8
Not completed — was arrested and put in jail | 0 | 1
Not completed — non study related adverse event | 1 | 0
Not completed — Blood Pressure outside study parameters | 2 | 0

BASELINE CHARACTERISTICS:
Population: Those eligible participants who received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Doxazosin | Placebo | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 7 | 5 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 6 | 7 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in Psychostimulant-positive Urines Over Time
Description: Urine samples positive for methamphetamine or cocaine via twice-weekly urine drug screens. Weekly urine results data were averaged within subjects and the mean proportion across subjects within each group was calculated for graphic representation.
Time Frame: twice-weekly urine samples (8 weeks)
Population: Those eligible participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: proportion of psychostimulant-pos urines
Units Other Than Participants: Urine samples
Arm/Group | Doxazosin | Placebo
Number analyzed (Participants) | 11 | 11
Number analyzed (Urine samples) | 89 | 77
proportion of psychostimulant-pos urines
  Week 1 (N=10, 11) | .6 (.52) | .41 (.49)
  Week 2 (N=7, 8) | .79 (.39) | .25 (.38)
  Week 3 (N=6, 5) | .58 (.49) | .4 (.55)
  Week 4 (N=6, 4) | .75 (.42) | .5 (.58)
  Week 5 (N=4, 4) | .5 (.41) | .25 (.29)
  Week 6 (N=4, 3) | .63 (.25) | 0 (0)
  Week 7 (N=4, 3) | 1 (0) | 0 (0)
  Week 8 (N=3, 2) | .83 (.29) | .25 (.35)
Statistical Analysis 1: Comparison: Doxazosin vs Placebo; The analysis was applied to urine data obtained at all time points during weeks 1-8; Test type: Superiority or Other; p = 0.05, Regression, Logistic; Odds Ratio (OR) = 1.0529

ADVERSE EVENTS:
Arm/Group | Doxazosin | Placebo
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/11
Other Adverse Events (participants affected / at risk) | 8/11 | 4/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxazosin (N=11) | Placebo (N=11)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxazosin (N=11) | Placebo (N=11)
Muscle Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Numbness in fingertips (Nervous system disorders) | 1 (1) | 0 (0)
nausea, abdominal cramps (Gastrointestinal disorders) | 1 (1) | 1 (1)
black eye (Eye disorders) | 1 (1) | 0 (0)
palpitations with shortness of breath (Psychiatric disorders) | 1 (1) | 0 (0)
Drowsiness, Fatigue (General disorders) | 1 (1) | 1 (1)
Sweating (General disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Head edema from fight (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sleep Disturbances (General disorders) | 1 (1) | 1 (1)
Elevated blood pressure (Cardiac disorders) | 2 (2) | 0 (0)
Abdominal pain and pain on urinating (Renal and urinary disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (Cardiac disorders) | 0 (0) | 1 (1)
Orthostatic Hypotension (Cardiac disorders) | 0 (0) | 1 (1)
Lightheadedness, dizziness (General disorders) | 1 (1) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No